CLINICAL TRIAL: NCT06932549
Title: Engaging Partners in Caring Communities
Acronym: EPICC
Status: Enrolling by invitation | Type: Observational
Sponsor: Tennessee State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #HS2021-4674
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Disease Prevention
Keywords: community-engaged research; health equity; health disparities; implementation science; faith-based organizations

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- There will be a single cohort consisting of up to 40 congregations.: The study cohort will consist of up to 40 congregations in Davidson County, TN that that have had a physical location for at least a year, have approval from their leader, and have a tax ID will be eligible for enrollment. Each will be offered up to 10 months of at least 1 hour/month of technical assistance for implementing an evidence-based (EB) chronic disease prevention congregation-level intervention selected by the congregation from five identified by the study team. The study team identified the five EB Programs through a systematic search of federal websites, selecting those programs that address chronic diseases that disproportionately affect African Americans, that can be delivered by non-health care providers in community settings. The selected programs include materials, including facilitator guidance, that are downloadable at no charge
  Interventions: Behavioral: Technical assistance is designed to integrate Expert Recommendations for Implementing Change (ERIC) strategies, and Getting To Outcomes-TA.

INTERVENTIONS:
Behavioral: Technical assistance is designed to integrate Expert Recommendations for Implementing Change (ERIC) strategies, and Getting To Outcomes-TA. — The TA is tailored to each congregation using the results of the implementation capacity survey completed by the congregation's team and materials from the EB Program selected by the congregation. The TA teams of two research staff are being trained and coached by Dr. Abe Wandersman, lead developer of Getting To Outcomes-TA (GTO-TA). TA sessions are audio-recorded and will be evaluated for fidelity to GTO-TA, and use of specific ERIC strategies.

SUMMARY:
The goal of the EPICC observational study is to learn about capacity to implement evidence-based health promotion programs (EBPs) in congregations that are offered semi-structured technical assistance (TA). Congregational teams will complete an implementation capacity assessment survey before the TA is offered and 10 months later, after TA has been provided for up to 10 months. Participating congregations will be a convenience sample of congregations in Davidson County, TN that serve primarily African American communities.

DETAILED DESCRIPTION:
The recruitment process is designed to provide a team of 3-5 volunteers from 40 congregations with information about five EBPs identified by the research team from which they are to choose one. The team completes one EPICC Survey for their congregation. The team is then offered up to 10 months of TA with the expectation that 2-3 months will be used for planning to launch the EBP, with 4-6 months for implementation. Each congregation will be asked to recruit a minimum of 8-10 members of the congregation to complete a brief report of health behaviors prior to launching of the EBP and repeating that report 6 months later to assess the impact of the EBP on their health behaviors.

ELIGIBILITY:
Inclusion Criteria: Adult (18 years and older) participants in the behavioral intervention (implemented health promotion program) in a congregation in Davidson County that has completed enrollment in the EPICC Project.

Exclusion Criteria:

* Individuals who are not enrolled in a health promotion program implemented in an EPICC congregation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected congregations are all in Davidson County, TN and self-identify as serving African Americans. The proportion of African Americans considered to be members of the congregation may fluctuate over time and will be estimated by church leaders. Some EB programs are designed to serve families and so there may be individuals participating in EB programs who are minors; however, no data will be obtained from minors.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Engaging Partners in Caring Communities (EPICC) Survey | Congregational teams complete the EPICC Survey at baseline and again 6-10 months later.
  The EPICC Survey was developed using the Consolidated Framework for Implementation Research (CFIR) and building on other surveys for measuring congregational readiness for health promotion. It consists of

SECONDARY OUTCOMES:
My Own Health Report | My Own Health Report will be completed when the congregation launches their health promotion program and again 6 months later.
  This is a brief self-reported screening of health-related behavior that will be completed in REDCap. It includes items related to frequency of consumption of fruits, vegetables, and sugary beverages, strenuous exercise, stress, tobacco and alcohol use over the previous 7 days. There are also items about transportation access, housing and food security. Each congregation will be asked to recruit 8-10 individuals who intend to participate in some aspect of the EB Program being implemented by the church. These individuals will be guided to create a unique ID number they can remember so that their reports are anonymous.

CONTACTS AND LOCATIONS:
Locations (1):
- Tennessee State University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss this with congregations that enroll in the study. They will be given the option of allowing or prohibiting sharing of individual data from My Own Health Report.

REFERENCES:
- See also: The EPICC website is an evolving source of information about the project, and will eventually include information from participating congregations that they ask to have shared. — https://theepiccproject.org/